CLINICAL TRIAL: NCT03767738
Title: A Study in Patients With Chorioretinal Vascular Disease to Evaluate an Aflibercept (EYLEA®) Prefilled Syringe
Brief Title: Study to Evaluate an Aflibercept (EYLEA®) Prefilled Syringe
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VGFTe-OD-1881
Record Dates: First submitted 2018-12-05; First posted 2018-12-07 (Actual); Results first posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-08

CONDITIONS: Chorioretinal Vascular Disease
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intravitreal Aflibercept Injection (IAI) (Experimental): Cohort 1 - Initial patients Cohort 2 - Additional patients
  Interventions: Drug: Intravitreal Aflibercept Injection (IAI)

INTERVENTIONS:
Drug: Intravitreal Aflibercept Injection (IAI) — IAI prepared and administered with a pre-filled syringe (PFS)
  Other Names: Aflibercept; EYLEA®

SUMMARY:
The primary objective of the study is to determine if the pre-filled syringe (PFS) supports successful preparation and accurate administration of an aflibercept injection.

The secondary objective of the study is to assess ocular safety in the study eye.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants who have neovascular age-related macular degeneration (AMD), diabetic macular edema (DME), retinal vein occlusion (RVO), or diabetic retinopathy (DR) with diabetic macular edema (DME) in the study eye

Key Exclusion Criteria:

* Evidence of active infectious blepharitis, keratitis, scleritis, or conjunctivitis in either eye
* Any active intraocular inflammation or infection in either eye or history of intraocular inflammation or infection after past intravitreal injection treatment (IVT) injections with any agent in either eye
* History of or any current indication of excessive bleeding and recurrent hemorrhages, including any prior excessive intraocular (including subconjunctival) bleeding or hemorrhages after IVT injection or intraocular procedures in either eye
* Any intraocular surgery in the study eye at any time during the past 3 months
* Current systemic infectious disease or a therapy for active infectious disease
* Pregnant or breastfeeding women

Note: Other inclusion/ exclusion apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2020-08-19 (Actual); Study Completion 2020-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (2):
- United States (2):
  - Regeneron Study Site, Houston, Texas
  - Regeneron Study Site, The Woodlands, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 65 participants were enrolled in the United States.
Units Other Than Participants: Eyes
Groups:
- Cohort 1: Intravitreal Aflibercept Injection (IAI) 2 mg: Participants in cohort 1 received a single IAI in a prefilled syringe (PFS) at a dose of 2 milligrams (mg) on Day 1.
- Cohort 2: IAI 2 mg: Participants in cohort 2 received a single IAI in a PFS at a dose of 2 mg on Day 1.
Period: Overall Study
Arm/Group | Cohort 1: Intravitreal Aflibercept Injection (IAI) 2 mg | Cohort 2: IAI 2 mg
Started | 35; 35 Eyes | 30; 30 Eyes
Completed | 35; 35 Eyes | 30; 30 Eyes
Not Completed | 0; 0 Eyes | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Intravitreal Aflibercept Injection (IAI) 2 mg | Cohort 2: IAI 2 mg | Total
Number analyzed (Participants) | 35 | 30 | 65
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.2 (10.04) | 64.7 (13.44) | 68.8 (12.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 14 | 34
  Male | 15 | 16 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 32 | 26 | 58
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants] — Race
  Participants
    White | 32 | 25 | 57
    Black or African American | 3 | 3 | 6
    Asian | 0 | 1 | 1
    American Indian or Alaska Native | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Other | 0 | 1 | 1
    Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Aflibercept Injections Successfully Administered Utilizing the Prefilled Syringe (PFS)
Description: Participants received a single dose of study drug, administered in the selected study eye with the PFS by a retina specialist. Physician assessed successful aflibercept preparation and administration with the PFS.
Time Frame: At Day 1
Population: Safety analysis set (SAF) included all enrolled participants who received study drug.
Measure: Number; unit: Injections
Arm/Group | Cohort 1: Intravitreal Aflibercept Injection (IAI) 2 mg | Cohort 2: IAI 2 mg
Number analyzed (Participants) | 35 | 30
Injections | 35 | 29

2. Secondary Outcome: Incidence of Ocular Treatment-Emergent Adverse Events (TEAEs) of Study Eye Through Day 29
Description: A treatment emergent AE (TEAE) is an adverse event starting after study eye injection and no later than 28 days after administration of study medication.
Time Frame: Baseline through Day 29
Population: SAF included all enrolled participants who received study drug.
Measure: Number; unit: Events
Units Other Than Participants: Eyes
Arm/Group | Cohort 1: Intravitreal Aflibercept Injection (IAI) 2 mg | Cohort 2: IAI 2 mg
Number analyzed (Participants) | 35 | 30
Number analyzed (Eyes) | 35 | 30
Events
  Conjunctival haemorrhage | 3 | 1
  Eye irritation | 3 | 0
  Dry eye | 0 | 1
  Eye pain | 0 | 1
  Lenticular opacities | 0 | 1
  Corneal abrasion | 1 | 0

3. Secondary Outcome: Incidence of Ocular Serious TEAEs of Study Eye Through Day 29
Description: A serious treatment emergent AE (TEAE) is a serious adverse event starting after study eye injection and no later than 28 days after administration of study medication.
Time Frame: Baseline through Day 29
Population: SAF included all enrolled participants who received study drug.
Measure: Number; unit: Events
Units Other Than Participants: Eyes
Arm/Group | Cohort 1: Intravitreal Aflibercept Injection (IAI) 2 mg | Cohort 2: IAI 2 mg
Number analyzed (Participants) | 35 | 30
Number analyzed (Eyes) | 35 | 30
Events | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Day 29
Arm/Group | Cohort 1: Intravitreal Aflibercept Injection (IAI) 2 mg | Cohort 2: IAI 2 mg
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/30
Serious Adverse Events (participants affected / at risk) | 1/35 | 0/30
Other Adverse Events (participants affected / at risk) | 6/35 | 1/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Intravitreal Aflibercept Injection (IAI) 2 mg (N=35) | Cohort 2: IAI 2 mg (N=30)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Intravitreal Aflibercept Injection (IAI) 2 mg (N=35) | Cohort 2: IAI 2 mg (N=30)
Conjunctival haemorrhage Study Eye (Eye disorders) | 3 (3) | 1 (1)
Eye irritation Study Eye (Eye disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2020-05-01): https://cdn.clinicaltrials.gov/large-docs/38/NCT03767738/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-06): https://cdn.clinicaltrials.gov/large-docs/38/NCT03767738/SAP_001.pdf